CLINICAL TRIAL: NCT05862350
Title: Effects of Lavender Essential Oil on Sleep Quality, Anxiety, and Fatigue in Patients With Chronic Heart Failure
Brief Title: Effects of Lavender Essential Oil in Patients With Chronic Heart Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2022LSK-400
Record Dates: First submitted 2022-10-24; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2022-10

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; lavender essential oil; sleep quality; Anxiety Disorders; Fatigue
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Fatigue | interventions — lavender oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy inhalation with lavender essential oil (Experimental): Patients in this group will receive aromatherapy inhalation with lavender essential oil for 28 days , and their sleep quality, anxiety and fatigue will be evaluated at baseline, the 7th day, and 28th day.
  Interventions: Other: aromatherapy inhalation with lavender essential oil
- Aromatherapy inhalation with coconut essential oil (Placebo Comparator): Patients in this group will receive aromatherapy inhalation with coconut essential oil for 28 days , and their sleep quality, anxiety and fatigue will be evaluated at baseline, the 7th day, and 28th day.
  Interventions: Other: aromatherapy inhalation with coconut essential oil.

INTERVENTIONS:
Other: aromatherapy inhalation with lavender essential oil — patients in the experimental group will receive aromatherapy inhalation by 4 drops of 50% lavender essential oil，which is diluted with coconut essential oil， on the cotton chip in the diffuser clip for 8 hours each night during sleep
  Arms: Aromatherapy inhalation with lavender essential oil
Other: aromatherapy inhalation with coconut essential oil. — patients in the experimental group will receive aromatherapy inhalation by 4 drops of 100% coconut essential oil on the cotton chip in the diffuser clip for 8 hours each night during sleep
  Arms: Aromatherapy inhalation with coconut essential oil

SUMMARY:
The goal of the trial is to study the effects of lavender essential oil on sleep quality, anxiety, and fatigue in patients with chronic heart failure. The main questions it may answer are

1. effects of lavender essential oil on sleep quality
2. effects of lavender essential oil on anxiety
3. effects of lavender essential oil on fatigue

Patients will be randomly divided into experimental and control groups, the control group will inhale essential coconut oil, and the experimental group will inhale lavender essential oil for four weeks. At baseline, on the 7th day, and 28th day, the sleep quality, anxiety, and fatigue will be evaluated.

DETAILED DESCRIPTION:
Heart failure (HF)， a severe manifestation or advanced stage of various cardiac diseases, may seriously affect patients' quality of life because repeated hospitalizations lead to changes in work and living environment, changes in roles, economic burdens, sexual dysfunction, limitations of social life, and worries about maintaining life. Patients are often accompanied by mental problems such as anxiety, depression, fatigue, and sleep disorders, so their quality of life is low.

Currently, the treatment of CHF is mainly to improve physical symptoms and control complications. However, insufficient attention is drawn to mental and psychological problems such as anxiety, sleep disorders, and fatigue associated with CHF patients.

Patients with anxiety and sleep disturbances are generally treated with antipsychotic and sedative-hypnotic drugs. Although effective, this method also creates dependencies and tolerability with the long-term application. So in recent years, complementary and alternative medicine is a novel adjunctive therapy, including aromatherapy, and traditional medicine, which can improve the patient's health and maintain a calm inner peace.

The commonly used lavender essential oil (Lavandula angustifolia) is the least toxic and allergenic of all aromatic oils. The main components of lavender are linalool and linalool acetate, which act as sedative, anti-nociceptive, and antispasmodic by reducing sympathetic nerve activity and stimulating the parasympathetic nervous system activity. Aromatherapy using lavender essential oil has been widely used in patients with cancer, postpartum depression, pregnant women, blood purification, acute coronary syndrome, myocardial infarction, and quasi-coronary angiography. Studies have shown that aromatherapy using lavender essential oil can relieve anxiety and depression, reduce fatigue, and improve sleep quality, and it has not been found to cause associated adverse events and complications. It showed good safety, while the use of lavender essential oil in patients with CHF has been less studied.

This study intends to use aromatherapy for CHF patients to observe the effects of lavender essential oil inhalation on sleep quality, anxiety, and fatigue in CHF patients, in order to provide a new care method for CHF patients with all-round mental and physical self-management and improve the long-term quality of life of CHF patients.

ELIGIBILITY:
Inclusion Criteria:

* Met the diagnostic criteria of heart failure:cardiac function grade ⅱ-ⅲ, disease duration ≥6 months.
* Blood pressure ≥90/60mmH, heart rate ≥60 times/min.
* No malignant arrhythmia, no need for oxygen or mechanical ventilation.
* Pittsburgh sleep quality (PSQI) score > 5, State-trait anxiety scale (STAI) score 21-59.
* No nasal diseases, normal sense of smell.
* Normal hearing and language expression, able to communicate, volunteer to participate in this study.

Exclusion Criteria:

* Pregnant women.
* Suffering from physical pain diseases or combined with tumors and other serious diseases of the system
* A history of mental illness, the use of psychiatric or sedative hypnotic drugs within 1 month.
* Allergic constitution, allergic to lavender essential oil or coconut oil, suffering from allergic rhinitis, eczema, asthma and other respiratory diseases.
* Declined to participate in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Change of Pittsburgh Sleep Quality Index | at base line,7th day, 14th day, 28th day
  The Pittsburgh Sleep Quality Index assesses sleep quality, with scores ranging from 0 to 21. Higher scores mean poorer sleep quality.
Change of State-trait anxiety inventory | at base line,7th day, 14th day, 28th day
  The State-trait anxiety inventory is used to assess state anxiety and trait anxiety on a scale from 20 to 80, with higher scores meaning more severe anxiety.
Change of the Fatigue Assessment Scale | at base line,7th day, 14th day, 28th day
  The Fatigue Assessment Scale assesses fatigue levels on a scale of 10 to 50, with higher scores meaning more fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Jingwen Hu, Master, Principal Investigator — the First Afiliated Hospital of Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drexler H, Coats AJ. Explaining fatigue in congestive heart failure. Annu Rev Med. 1996;47:241-56. doi: 10.1146/annurev.med.47.1.241. PMID 8712779
- [Background] Easton K, Coventry P, Lovell K, Carter LA, Deaton C. Prevalence and Measurement of Anxiety in Samples of Patients With Heart Failure: Meta-analysis. J Cardiovasc Nurs. 2016 Jul-Aug;31(4):367-79. doi: 10.1097/JCN.0000000000000265. PMID 25930162
- [Background] Kessing D, Denollet J, Widdershoven J, Kupper N. Fatigue and self-care in patients with chronic heart failure. Eur J Cardiovasc Nurs. 2016 Aug;15(5):337-44. doi: 10.1177/1474515115575834. Epub 2015 Feb 25. PMID 25715645
- [Background] Steinhorn DM, Din J, Johnson A. Healing, spirituality and integrative medicine. Ann Palliat Med. 2017 Jul;6(3):237-247. doi: 10.21037/apm.2017.05.01. Epub 2017 May 22. PMID 28595441
- [Background] Cavanagh HM, Wilkinson JM. Biological activities of lavender essential oil. Phytother Res. 2002 Jun;16(4):301-8. doi: 10.1002/ptr.1103. PMID 12112282
- [Background] Cheraghbeigi N, Modarresi M, Rezaei M, Khatony A. Comparing the effects of massage and aromatherapy massage with lavender oil on sleep quality of cardiac patients: A randomized controlled trial. Complement Ther Clin Pract. 2019 May;35:253-258. doi: 10.1016/j.ctcp.2019.03.005. Epub 2019 Mar 8. PMID 31003666
- [Background] Dos Reis Lucena L, Dos Santos-Junior JG, Tufik S, Hachul H. Lavender essential oil on postmenopausal women with insomnia: Double-blind randomized trial. Complement Ther Med. 2021 Jun;59:102726. doi: 10.1016/j.ctim.2021.102726. Epub 2021 Apr 24. PMID 33905827
- [Background] Lee J, Hur MH. The Effects of Aroma Essential Oil Inhalation on Stress, Pain, and Sleep Quality in Laparoscopic Cholecystectomy Patients: A Randomized Controlled Trial. Asian Nurs Res (Korean Soc Nurs Sci). 2022 Feb;16(1):1-8. doi: 10.1016/j.anr.2021.11.002. Epub 2021 Dec 24. PMID 34954406
- [Background] Shammas RL, Marks CE, Broadwater G, Le E, Glener AD, Sergesketter AR, Cason RW, Rezak KM, Phillips BT, Hollenbeck ST. The Effect of Lavender Oil on Perioperative Pain, Anxiety, Depression, and Sleep after Microvascular Breast Reconstruction: A Prospective, Single-Blinded, Randomized, Controlled Trial. J Reconstr Microsurg. 2021 Jul;37(6):530-540. doi: 10.1055/s-0041-1724465. Epub 2021 Feb 6. PMID 33548936
- [Background] Moradi K, Ashtarian H, Danzima NY, Saeedi H, Bijan B, Akbari F, Mohammadi MM. Essential Oil from Citrus aurantium Alleviates Anxiety of Patients Undergoing Coronary Angiography: A Single-Blind, Randomized Controlled Trial. Chin J Integr Med. 2021 Mar;27(3):177-182. doi: 10.1007/s11655-020-3266-5. Epub 2020 Jun 22. PMID 32572778
- [Derived] Hu J, Chong MS, Jia Y, Wu Y, Li J, Wang W. Effects of lavender essential oil inhalation on sleep quality and fatigue in patients with chronic heart failure: a randomised controlled trial. Eur J Cardiovasc Nurs. 2026 Jan 7:zvag006. doi: 10.1093/eurjcn/zvag006. Online ahead of print. PMID 41499426